CLINICAL TRIAL: NCT06047210
Title: An Observational, Multicenter Study to Evaluate Levels of Interferon Gamma (IFNγ) and Other Inflammatory Mediators in Adult Patients With Hemophagocytic Lymphohistiocytosis (A-HLH)
Brief Title: Evaluation of IFNγ and Inflammatory Mediators in Patients With Hemophagocytic Lymphohistiocytosis
Status: Completed | Type: Observational
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: Brigham and Women's Hospital (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Sponsor
Other Study IDs: NI-0501-08
Record Dates: First submitted 2023-08-25; First posted 2023-09-21 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Hemophagocytic Lymphohistiocytoses
Keywords: Hemophagocytic Lymphohistiocytosis; Interferon Gamma; IFNγ; Biomarkers; Inflammatory Markers
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — For biomarker analysis a maximum of 5 milliliter (mL) of whole blood was required per time point.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A-HLH Patients: Patients diagnosed with A-HLH.
  Interventions: Other: Blood Draws Data Collection
- Malignancy-Associated Hemophagocytic Lymphohistiocytosis (M-HLH) Patients: Patients diagnosed with HLH in the context of a malignancy.
  Interventions: Other: Blood Draws Data Collection

INTERVENTIONS:
Other: Blood Draws Data Collection

SUMMARY:
This observational study is designed to provide a better understanding of the potential use of interferon gamma (IFNγ) and IFNγ-inducible chemokines as markers of HLH disease activity in adults, and the potential of IFNγ to represent a therapeutic target.

DETAILED DESCRIPTION:
This is a observational study designed to determine the levels of pro-inflammatory markers in adult patients diagnosed with HLH and to assess the relationship between the biomarkers and disease activity in these patients during the HLH course. Inflammatory markers include IFNγ and IFNγ-induced chemokines C-X-C chemokine ligand 9 and C-X-C chemokine ligand 10.

In addition to the blood samples for the biomarker analysis, relevant information gathered by the treating physician will be collected in a data collection form. Whenever possible, collection of serum samples for biomarker analysis and relevant information should occur at HLH diagnosis, at regular time intervals during the treatment course (not more than once a week) up to resolution of HLH.

Blood samples will also be sent to the study sponsor (NovImmune S.A.) for cytokine testing. Before patient's samples are sent to the sponsor for testing, patient's name and any personal identifying information will be coded to protect participant's privacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients >=18 years old diagnosed with active HLH as established by the treating physician.
* HLH forms of unknown origin or secondary to infections or rheumatologic disorders.
* Should the diagnosis of primary HLH or malignancy become apparent after inclusion, the data collected will be analyzed separately as additional cohorts.
* The patient must have consented to the use of their clinical data for research purposes at the site.

Exclusion Criteria:

* Patients with primary HLH (diagnosed by the presence of homozygous mutations in a known HLH causative gene) and secondary HLH due to malignancy are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female adult (>=18 years old) patients who are diagnosed with HLH and meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Berliner, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Brigham and Women's Hospital — https://www.brighamandwomens.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 4 observational study was conducted in adult patients diagnosed with hemophagocytic lymphohistiocytosis (A-HLH) at a single center in the United States of America.
Pre-assignment Details: A total of 14 patients were enrolled in the study.
Period: Overall Study
Arm/Group | A-HLH Patients | Malignancy-Associated Hemophagocytic Lymphohistiocytosis (M-HLH) Patients
Started | 10 | 4
Completed | 10 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The enrolled set included all patients who signed an informed consent.
Groups:
- M-HLH Patients: Patients diagnosed with HLH in the context of a malignancy.
- Total: Total of all reporting groups
Arm/Group | A-HLH Patients | M-HLH Patients | Total
Number analyzed (Participants) | 10 | 4 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (12.4) | 54.3 (4.9) | 47.5 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 6 | 2 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 8 | 3 | 11
  African descent | 1 | 0 | 1
  Mixed/multi-racial | 1 | 0 | 1
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Serum Concentration of Inflammatory Biomarker - C-X-C Chemokine Ligand 10 (CXCL10)
Description: Serum samples was collected at various times after HLH diagnosis to determine the concentration of CXCL10.
Time Frame: 11 months
Population: The enrolled set included all patients who signed an informed consent. Only patients with data collected for this outcome measure are reported.
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/mL)
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 9 | 2
picogram/milliliter (pg/mL) | 2079.286 (2659.228) | 15197.143 (21288.948)

2. Primary Outcome: Mean Serum Concentration of Inflammatory Biomarker - C-X-C Chemokine Ligand 9 (CXCL9)
Description: Serum samples was collected at various times after HLH diagnosis to determine the concentration of CXCL9.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 9 | 2
pg/mL | 4474.685 (10207.638) | 6602.853 (7777.846)

3. Primary Outcome: Mean Serum Concentration of Inflammatory Biomarker - Interferon Gamma (IFNg)
Description: Serum samples was collected at various times after HLH diagnosis to determine the concentration of IFNg.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 9 | 2
pg/mL | 81.782 (140.870) | 809.810 (769.433)

4. Primary Outcome: Mean Serum Concentration of Inflammatory Biomarker - Interleukin 10 (IL-10)
Description: Serum samples was collected at various times after HLH diagnosis to determine the concentration of IL-10.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 9 | 2
pg/mL | 24.157 (87.640) | 266.948 (257.770)

5. Primary Outcome: Mean Serum Concentration of Inflammatory Biomarker - Interleukin 1 Beta (IL-1B)
Description: Serum samples was collected at various times after HLH diagnosis to determine the concentration of IL-1B.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 9 | 2
pg/mL | 2.140 (0.000) | 2.140 (0.000)

6. Primary Outcome: Mean Serum Concentration of Inflammatory Biomarker - Interleukin 6 (IL-6)
Description: Serum samples was collected at various times after HLH diagnosis to determine the concentration of IL-6.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 9 | 2
pg/mL | 3.455 (3.727) | 29.695 (52.403)

7. Primary Outcome: Mean Serum Concentration of Inflammatory Biomarker - Neopterin
Description: Serum samples was collected at various times after HLH diagnosis to determine the concentration of neopterin.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanomoles
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 9 | 2
nanomoles | 33.995 (29.227) | 839.775 (950.070)

8. Primary Outcome: Mean Serum Concentration of Inflammatory Biomarker - Tumor Necrosis Factor Alpha (TNFa)
Description: Serum samples was collected at various times after HLH diagnosis to determine the concentration of TNFa.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 9 | 2
pg/mL | 6.050 (6.405) | 14.308 (12.010)

9. Primary Outcome: Mean Serum Concentration of Inflammatory Biomarker - Total Human Interferon Gamma (hIFNg)
Description: Serum samples was collected at various times after HLH diagnosis to determine the concentration of hIFNg.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 9 | 2
pg/mL | 34.178 (25.950) | 1069.215 (1987.409)

10. Primary Outcome: Mean Serum Concentration of Inflammatory Biomarker - Soluble CD163 (sCD163)
Description: Serum samples was collected at various times after HLH diagnosis to determine the concentration of sCD163.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanogram (ng)/mL
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 4 | 1
nanogram (ng)/mL | 1431.488 (1078.058) | 878.880 (NA) — Standard deviation could not be determined when only 1 patient analyzed.

11. Primary Outcome: Mean Serum Concentration of Inflammatory Biomarker - Soluble IL-2 Receptor Alpha (sIL2Ra)
Description: Serum samples was collected at various times after HLH diagnosis to determine the concentration of sIL2Ra.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 9 | 2
pg/mL | 2273.193 (2383.154) | 27052.498 (24009.516)

12. Primary Outcome: Mean Serum Concentration of White Blood Cells
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of white blood cells.
Time Frame: 11 months
Population: The enrolled set included all patients who signed an informed consent.
Measure: Mean (Standard Deviation); unit: cells*10^3/microliter (mcL)
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 10 | 4
cells*10^3/microliter (mcL) | 4.263 (3.480) | 2.459 (2.854)

13. Primary Outcome: Mean Serum Concentration of Red Blood Cells
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of red blood cells.
Time Frame: 11 months
Population: The enrolled set included all patients who signed an informed consent.
Measure: Mean (Standard Deviation); unit: cells*10^6/mcL
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 10 | 4
cells*10^6/mcL | 3.420 (0.745) | 3.206 (0.396)

14. Primary Outcome: Mean Serum Concentration of Hemoglobin
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of hemoglobin.
Time Frame: 11 months
Population: The enrolled set included all patients who signed an informed consent.
Measure: Mean (Standard Deviation); unit: gram/deciliter (g/dL)
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 10 | 4
gram/deciliter (g/dL) | 10.11 (1.93) | 9.83 (1.09)

15. Primary Outcome: Mean Serum Concentration of Hematocrit
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of hematocrit.
Time Frame: 11 months
Population: The enrolled set included all patients who signed an informed consent.
Measure: Mean (Standard Deviation); unit: percentage of volume of red cells
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 10 | 4
percentage of volume of red cells | 30.03 (5.75) | 28.55 (3.55)

16. Primary Outcome: Mean Serum Concentration of Platelets
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of platelets.
Time Frame: 11 months
Population: The enrolled set included all patients who signed an informed consent.
Measure: Mean (Standard Deviation); unit: cells*10^3/mcL
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 10 | 4
cells*10^3/mcL | 182.6 (138.2) | 92.9 (87.1)

17. Primary Outcome: Mean Serum Concentration of Neutrophils
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of neutrophils.
Time Frame: 11 months
Population: The enrolled set included all patients who signed an informed consent.
Measure: Mean (Standard Deviation); unit: cells*10^3/mcL
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 10 | 4
cells*10^3/mcL | 7.715 (14.003) | 22.303 (37.944)

18. Primary Outcome: Mean Serum Concentration of Lymphocytes
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of lymphocytes.
Time Frame: 11 months
Population: The enrolled set included all patients who signed an informed consent.
Measure: Mean (Standard Deviation); unit: cells*10^3/mcL
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 10 | 4
cells*10^3/mcL | 3.636 (10.880) | 1.956 (3.424)

19. Primary Outcome: Mean Serum Concentration of Monocytes
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of monocytes.
Time Frame: 11 months
Population: The enrolled set included all patients who signed an informed consent.
Measure: Mean (Standard Deviation); unit: cells*10^3/mcL
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 10 | 4
cells*10^3/mcL | 1.306 (3.602) | 0.948 (1.721)

20. Primary Outcome: Mean Serum Concentration of Eosinophils
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of eosinophils.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells*10^3/mcL
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 9 | 4
cells*10^3/mcL | 0.252 (0.707) | 1.002 (2.449)

21. Primary Outcome: Mean Serum Concentration of Basophils
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of basophils.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells*10^3/mcL
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 9 | 4
cells*10^3/mcL | 0.181 (0.516) | 0.222 (0.399)

22. Primary Outcome: Mean Plasma Concentration of D-Dimer
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of D-dimer.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microgram (mcg)/mL
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 1 | 0
microgram (mcg)/mL | 2300.0 (NA) — Standard deviation could not be determined when only 1 patient analyzed. |

23. Primary Outcome: Mean Plasma Concentration of Fibrinogen
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of fibrinogen.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligram (mg)/dL
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 4 | 2
milligram (mg)/dL | 306.8 (145.7) | 172.5 (83.0)

24. Primary Outcome: Mean Activated Partial Thromboplastin Time (aPTT)
Description: Blood samples was collected at various times after HLH diagnosis to determine the aPTT.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 3 | 0
seconds | 27.98 (8.21) |

25. Primary Outcome: Mean Prothrombin Time
Description: Blood samples was collected at various times after HLH diagnosis to determine the prothrombin time.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 6 | 3
seconds | 13.81 (0.90) | 16.75 (4.60)

26. Primary Outcome: Mean Serum Concentration of C-Reactive Protein
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of c-reactive protein.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 5 | 3
mg/dL | 27.97 (31.13) | 13.35 (12.06)

27. Primary Outcome: Mean Serum Concentration of Ferritin
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of ferritin.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 9 | 3
ng/mL | 5050.2273 (5302.9183) | 24331.4517 (38189.6158)

28. Primary Outcome: Mean Plasma Concentration of Blood Urea Nitrogen
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of blood urea nitrogen.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 9 | 2
mg/dL | 17.3 (8.3) | 50.2 (37.3)

29. Primary Outcome: Mean Serum Concentration of Creatinine
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of creatinine.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 9 | 4
mg/dL | 0.768 (0.293) | 1.449 (0.748)

30. Primary Outcome: Mean Serum Concentration of Albumin
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of albumin.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gram/dL
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 9 | 4
gram/dL | 3.68 (0.55) | 3.21 (0.87)

31. Primary Outcome: Mean Serum Concentration of Sodium
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of sodium.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimoles/L
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 9 | 4
millimoles/L | 136.4 (3.7) | 135.3 (3.2)

32. Primary Outcome: Mean Serum Concentration of Fasting Triglycerides
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of fasting triglycerides.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 0 | 1
mg/dL |  | 645.0 (NA) — Standard deviation could not be determined when only 1 patient analyzed.

33. Primary Outcome: Mean Serum Concentration of Total Bilirubin
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of total bilirubin.
Time Frame: 11 months
Population: The enrolled set included all patients who signed an informed consent.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 10 | 4
mg/dL | 0.590 (0.559) | 4.204 (6.359)

34. Primary Outcome: Mean Serum Concentration of Conjugated Bilirubin
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of conjugated bilirubin.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Units Other Than Participants: Samples
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 6 | 1
Number analyzed (Samples) | 8 | 2
mg/dL | 0.25 (0.31) | 12.80 (1.13)

35. Primary Outcome: Mean Serum Concentration of Alanine Aminotransferase
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of alanine aminotransferase.
Time Frame: 11 months
Population: The enrolled set included all patients who signed an informed consent.
Measure: Mean (Standard Deviation); unit: international units (IU)/L
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 10 | 4
international units (IU)/L | 93.2 (145.6) | 54.8 (35.1)

36. Primary Outcome: Mean Serum Concentration of Aspartate Aminotransferase
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of aspartate aminotransferase.
Time Frame: 11 months
Population: The enrolled set included all patients who signed an informed consent.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 10 | 4
IU/L | 66.0 (105.8) | 48.6 (35.4)

37. Primary Outcome: Mean Serum Concentration of Alkaline Phosphatase
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of alkaline phosphatase.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 9 | 2
IU/L | 121.1 (98.8) | 258.2 (188.5)

38. Primary Outcome: Mean Serum Concentration of Lactate Dehydrogenase
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of lactate dehydrogenase.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 9 | 3
IU/L | 539.8 (660.8) | 362.7 (274.4)

39. Primary Outcome: Mean Serum Concentration of Immunoglobulin G (IgG)
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of IgG.
Time Frame: 11 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | A-HLH Patients | M-HLH Patients
Number analyzed (Participants) | 5 | 1
mg/dL | 763.6 (579.3) | 996.0 (NA) — Standard deviation could not be determined when only 1 patient analyzed.

ADVERSE EVENTS:
Description: Adverse events collection is not applicable as this is an observational study. Safety analysis including all-cause mortality, serious adverse events and other (non-serious) adverse events were not monitored.
Arm/Group | A-HLH Patients | M-HLH Patients
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/10/NCT06047210/Prot_002.pdf
  • Statistical Analysis Plan (2021-05-31): https://cdn.clinicaltrials.gov/large-docs/10/NCT06047210/SAP_001.pdf